CLINICAL TRIAL: NCT00031681
Title: A Phase I Study of UCN-01 in Combination With Irinotecan in Resistant Solid Tumor Malignancies (Part I) and in Triple Negative (ER-Negative, PgR-Negative, HER-2 Not-Amplified) Recurrent Breast Cancers (Part II)
Brief Title: 7-Hydroxystaurosporine and Irinotecan Hydrochloride in Treating Patients With Metastatic or Unresectable Solid Tumors or Triple Negative Breast Cancer (Currently Accruing Only Triple-negative Breast Cancer Patients Since 6/8/2007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Washington University Siteman Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00019; NCI-2009-00019 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5582; WUSM-SCC-0102; CDR0000069215; UVACC-SCC-0102; SCC 01-02 (Other: University of Virginia); 5582 (Other: CTEP); P30CA044579 (NIH)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Advanced Adult Primary Liver Cancer; Carcinoma of the Appendix; Estrogen Receptor-negative Breast Cancer; Extensive Stage Small Cell Lung Cancer; Gastrointestinal Stromal Tumor; HER2-negative Breast Cancer; Metastatic Gastrointestinal Carcinoid Tumor; Ovarian Sarcoma; Ovarian Stromal Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adult Primary Liver Cancer; Recurrent Anal Cancer; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Borderline Ovarian Surface Epithelial-stromal Tumor; Recurrent Breast Cancer; Recurrent Cervical Cancer; Recurrent Colon Cancer; Recurrent Endometrial Carcinoma; Recurrent Esophageal Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Recurrent Gastric Cancer; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Cancer; Recurrent Prostate Cancer; Recurrent Rectal Cancer; Recurrent Salivary Gland Cancer; Recurrent Small Cell Lung Cancer; Recurrent Small Intestine Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Small Intestine Adenocarcinoma; Small Intestine Leiomyosarcoma; Small Intestine Lymphoma; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Anal Cancer; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Borderline Ovarian Surface Epithelial-stromal Tumor; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Endometrial Carcinoma; Stage IV Esophageal Cancer; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Gastric Cancer; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer; Stage IV Prostate Cancer; Stage IV Rectal Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer; Triple-negative Breast Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer; Unspecified Adult Solid Tumor, Protocol Specific; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Appendiceal Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Anus Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Esthesioneuroblastoma, Olfactory; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Salivary Gland Neoplasms; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms | interventions — 7-hydroxystaurosporine; Irinotecan

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): PART I: Patients receive irinotecan hydrochloride IV over 90 minutes on days 1, 8, 15, and 22 and 7-hydroxystaurosporine IV over 3 hours on days 2 and 23. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan hydrochloride and 7-hydroxystaurosporine until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Blood samples are collected periodically during study treatment.
  PART II: (treatment of triple negative recurrent breast cancer): Patients receive irinotecan hydrochloride IV and 7-hydroxystaurosporine IV as in part I at the MTD and undergo blood sample collection.
  Interventions: Drug: 7-hydroxystaurosporine; Drug: irinotecan hydrochloride; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Drug: 7-hydroxystaurosporine — Given IV
  Other Names: UCN-01
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving 7-hydroxystaurosporine together with irinotecan hydrochloride in treating patients with metastatic or unresectable solid tumors, including triple-negative breast cancer (currently enrolling only patients with triple-negative breast cancer since 6/8/2007). Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving 7-hydroxystaurosporine together with irinotecan hydrochloride may help kill more cancer cells by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of UCN-01 (7-hydroxystaurosporine) and irinotecan (irinotecan hydrochloride) in patients with resistant solid tumors. (Part I [closed to accrual as of 6/8/2007]) II. Determine the dose-limiting toxicity of this regimen in these patients. (Part I [closed to accrual as of 6/8/2007]) III. Determine the types of toxic effects of this regimen in these patients. (Part I [closed to accrual as of 6/8/2007]) IV. Determine the anti-tumor activity in terms of overall response rate (partial response [PR] and complete response [CR]), clinical benefit rate (PR, CR, and stable disease), and time to disease progression in patients with estrogen receptor-negative, progesterone receptor-negative, and HER-2 not amplified (triple negative) locally recurrent or metastatic breast cancer treated with this regimen. (Part II) V. Determine the side effect profile of this regimen in patients with triple negative recurrent breast cancer. (Part II)

SECONDARY OBJECTIVES:

I. Determine any anti-tumor activity of this regimen in these patients. (Part I [closed to accrual as of 6/8/2007]) II. Determine the pharmacokinetics of this regimen in these patients. (Part I [closed to accrual as of 6/8/2007]) III. Determine the activity of the serum α-acid glycoprotein and correlate this level with free UCN-01 concentrations. (Part I [closed to accrual as of 6/8/2007]) IV. Determine the in vivo mechanisms of UCN-01 activity in these patients.

OUTLINE: This is a dose-escalation study.

PART I: Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1, 8, 15, and 22 and 7-hydroxystaurosporine IV over 3 hours on days 2 and 23. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan hydrochloride and 7-hydroxystaurosporine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Blood samples are collected periodically during study treatment.

PART II: (treatment of triple negative recurrent breast cancer): Patients receive irinotecan hydrochloride IV and 7-hydroxystaurosporine IV as in part I at the MTD and undergo blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Part I (closed to accrual as of 6/8/2007)

  * Histologically confirmed solid tumor that is metastatic or unresectable for which standard curative measures do not exist or are no longer effective, including the following:

    * Gastrointestinal tract cancer
    * Lung cancer
    * Breast cancer
    * Ovarian cancer
    * Endometrial cancer
    * Cervical cancer
    * Prostate cancer
    * Head and neck cancer
  * Patients with or without measurable or evaluable disease allowed

    * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques or ≥ 10 mm with spiral CT scan

      * Tumor markers allowed for evaluable disease
      * Positive bone scan, osteoblastic metastases, and pleural or peritoneal effusions are not considered measurable or evaluable disease
  * No known brain metastases
* Part II

  * Histologically confirmed (either primary or the recurrent site) locally recurrent or metastatic breast cancer not amendable to surgery

    * Measurable disease

      * For skin lesions, documentation by color photography and estimation of lesion size with a ruler are required
  * Must have undergone prior therapy with an anthracycline and a taxane either in the adjuvant or metastatic setting
  * CNS metastasis allowed provided stable disease (i.e., no evidence of local progression) ≥ 3 months after local therapy
  * Hormone receptor status:

    * Estrogen receptor negative
    * Progesterone receptor negative
    * HER-2 not amplified by fluorescence in situ hybridization
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST/ALT no greater than 3 times upper limit of normal (ULN)
* No Gilbert's disease
* No chronic unconjugated hyperbilirubinemia
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min
* No symptomatic cardiac dysfunction
* No symptomatic pulmonary dysfunction
* Oxygen saturation at least 90% by pulse oximetry on room air at rest and after walking 6 minutes
* No insulin-dependent diabetes mellitus
* No other uncontrolled concurrent illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study entry
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to UCN-01 or irinotecan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent granulocyte colony-stimulating factors (filgrastim [G-CSF] or sargramostim [GM-CSF]) during the first course of study
* See Disease Characteristics (Part II)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior irinotecan allowed
* Less than 4 prior chemotherapy regimens in the adjuvant and/or metastatic setting (Part II)
* More than 4 weeks since prior radiotherapy and recovered
* Concurrent warfarin allowed
* Concurrent subcutaneous heparin allowed
* No other concurrent investigational agents
* No concurrent anticonvulsants (e.g., carbamazepine, phenobarbital, or phenytoin)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-12; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
MTD of irinotecan hydrochloride in combination with 7-hydroxystaurosporine in patients with resistant solid tumor malignancies (Part I) | Part I
  Defined as the highest dose given to at least 6 patients in which =< 1 out of 6 experience dose limiting toxicity (DLT).
DLT of irinotecan hydrochloride in combination with 7-hydroxystaurosporine in patients with resistant solid tumor malignancies (Part I) | Part I
Toxicities associated with irinotecan hydrochloride in combination with 7-hydroxystaurosporine in patients with resistant solid tumor malignancies (Part I) | Continuously over study treatment
  Graded using the Cancer Therapy Evaluation Program (CTEP) Active Version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Anti-tumor activity of 7-hydroxystaurosporine in combination with irinotecan hydrochloride in ER-negative, PgR-negative, HER-2 not-amplified (triple negative) recurrent breast cancer (Part II) | Every 6 weeks
  Including overall response rate (partial response [PR] +complete response [CR]), clinical benefit rate (PR+CR+stable disease [SD]), and time to disease progression. 95% confidence interval will be calculated. Evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Side effect profile of 7-hydroxystaurosporine in combination with irinotecan hydrochloride in triple negative recurrent breast cancer (Part II) | Continuously over study treatment
  95 % confidence interval will be calculated.

SECONDARY OUTCOMES:
Anti-tumor activity of the combination of irinotecan hydrochloride and 7-hydroxystaurosporine in treatment of patients with resistant solid tumor malignancies | Every 6 weeks
  Evaluated by the RECIST criteria.
Pharmacokinetics of irinotecan hydrochloride and 7-hydroxystaurosporine when administered in combination | Weekly during the first 4 weeks of course 1
  Using the high-performance liquid chromatography (HPLC) assays.
Serum alpha-acid glycoprotein and correlate this level with free 7-hydroxystaurosporine concentrations | Weekly during the first 4 weeks of course 1
In vivo mechanistic basis for 7-hydroxystaurosporine activity | Weekly during the first 4 weeks of course 1
  Explored by subgroup analysis (responders versus non-responders) on pharmacodynamic measures.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fracasso, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States